CLINICAL TRIAL: NCT02016404
Title: The Effect of a Low Sodium-High Potassium Salt on Blood Pressure in Vietnamese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: National Institute of Nutrition, Vietnam (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0793
Record Dates: First submitted 2013-12-09; First posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Hypertension
Keywords: blood pressure; sodium; salt; low sodium high potassium salt; potassium; Vietnam; randomized controlled trial
MeSH Terms: conditions — Hypertension | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-sodium, high-potassium salt (Active Comparator): Iodized low-sodium, high-potassium botcanh (a traditional mixture of salt, mono sodium glutamate (MSG), sugar and herbs) plus and iodized low-sodium, high-potassium salt for home food preparation
  Interventions: Other: Low-sodium, high-potassium salt
- Regular salt (Placebo Comparator): Regular iodized high-sodium botcanh (a traditional mixture of salt, MSG, sugar and herbs) and high-sodium salt
  Interventions: Other: Regular salt

INTERVENTIONS:
Other: Low-sodium, high-potassium salt — Iodized low-sodium, high-potassium botcanh (a traditional mixture of salt, MSG, sugar and herbs) plus and iodized low-sodium, high-potassium salt for home food preparation
  Arms: Low-sodium, high-potassium salt
Other: Regular salt — Regular iodized high-sodium botcanh (a traditional mixture of salt, MSG, sugar and herbs) and high-sodium salt
  Arms: Regular salt

SUMMARY:
The purpose of this study was to investigate the effects of low-sodium, high-potassium condiments and salt on blood pressure in untreated (pre)hypertensive Vietnamese adults.

ELIGIBILITY:
Inclusion Criteria:

Untreated prehypertension or mild hypertension (systolic BP between 130 and 160 mmHg and/or diastolic BP between 85 and 100 mmHg) based on the mean of two measurements with a 1-week interval

Exclusion Criteria:

Diagnosed or self-reported cardiovascular disease Diagnosed or self-reported kidney disease

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in office systolic blood pressure (SBP) | Change during 8 weeks of intervention
  Based on repeated measurements with a digital BP device (OMRONHEM 762) using the standard protocol of WHO STEP guideline at week 0, 2, 4 6 and 8.

SECONDARY OUTCOMES:
Change in office diastolic blood pressure (DBP) | Change during 8 weeks of intervention
  Based on repeated measurements with a digital BP device (OMRONHEM 762) using the standard protocol of WHO STEP guideline at week 0, 2, 4, 6 and 8.

OTHER OUTCOMES:
Change in 24-hour urinary sodium excretion | Change during 8 weeks of intervention
Change in 24-hour urinary potassium excretion | Change during 8 weeks of intervention
Change in body weight | Change during 8 weeks of intervention
Change in 24-hour urinary calcium excretion | Change during 8 weeks of intervention
Change in 24-hour urinary iodine excretion | Change during 8 weeks of intervention
Change in 24-hour urinary creatinine excretion | Change during 8 weeks of intervention
Change in 24-hour urinary protein | Change during 8 weeks of intervention
Change in heart rate | Change during 8 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ha TP Do, Principal Investigator — Community Nutrition, National Institute of Nutrition, Vietnam
Locations (1):
- National Institute of Nutrition (NIN), Department of Community Nutrition, Hanoi, Hai Ba Trung Dist., Vietnam

REFERENCES:
- See also: National Institute of Nutrition (NIN), Vietnam — http://viendinhduong.vn/home/en/Default.aspx